CLINICAL TRIAL: NCT02987374
Title: Pilot Study in Young Adults to Examine the Kinetics of Changes in the B-cell Repertoire Following TIV Immunization
Acronym: SLVP023
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Professor, Pediatrics, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SU-24167; U19AI057229-06 (NIH)
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Results first posted 2016-12-26 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Influenza
Keywords: Influenza Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2011-2012 Fluzone IIV3 (IM) (Other): Seasonal trivalent flu vaccine: NDC No 49281-011-50
  Interventions: Biological: 2011-2012 Fluzone IIV3 (IM)

INTERVENTIONS:
Biological: 2011-2012 Fluzone IIV3 (IM) — 2011-2012 Fluzone IIV3 vaccine delivered intramuscularly (IM)

SUMMARY:
The purpose is to investigate B-cell response to the trivalent Influenza Vaccine (TIV) in healthy young adults by vaccinating participants and obtaining blood samples at designated time points before and after vaccination.

DETAILED DESCRIPTION:
This is an exploratory study using a strategy that has not been previously employed to investigate B-cell responses. Investigators will collect blood samples from the volunteers at a higher frequency than in the two previous flu seasons to better define the dynamic response to vaccination. The objective is to compare the Ig gene repertoire before and after vaccination by deep sequencing PBMC and proteomic analysis of antibody CDR3 regions at 10 different time points before and after immunization.

This is a Phase IV study of healthy adults who are given standard TIV off-season. There are no exclusions for gender, ethnicity or race. Following confirmation of written informed consent, baseline blood samples will be drawn from all study participants at Day -5, Day -3 and Day 0 prior to immunization, and at Days 1, 4, 7, 9, 11, 28 and 180 post-immunization. Volunteers will be vaccine-naïve for the 2010-2011 and 2011-2012 seasonal influenza vaccines. All participants will receive a single dose of the current seasonal influenza vaccine by intramuscular (IM) injection at Day 0.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy, 18-30 year old young adult.
2. Availability for follow-up for the planned duration of the study at least 180 days after immunization.
3. Acceptable medical history by medical history and vital signs.

Exclusion Criteria:

1. Prior vaccination with 2010-2011 seasonal TIV or LAIV.
2. Prior off-study vaccination with the current 2011-2012 seasonal TIV or LAIV
3. Weight less than 110 pounds.
4. Allergy to egg or egg products, or to vaccine components, including gelatin or thimerosal (thimerosal in TIV multidose vials only).
5. Life-threatening reactions to previous influenza vaccinations
6. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
7. History of immunodeficiency (including HIV infection)
8. Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease, or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
9. Blood pressure >150 systolic or >95 diastolic at first study visit
10. Hospitalization in the past year for congestive heart failure or emphysema.
11. Chronic Hepatitis B or C.
12. Recent or current use of immunosuppressive medication, including systemic glucocorticoids. Corticosteroid nasal sprays and topical steroids are permissible.
13. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
14. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
15. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year.
16. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg. per day), Plavix, or Aggrenox must be reviewed by investigator to determine if this would affect the volunteer's safety.
17. Receipt of blood or blood products within the past 6 months.
18. Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
19. Receipt of inactivated vaccine 14 days prior to study enrollment, planned vaccinations prior to completion of Visit 09 (Day 28 after study vaccination), or planned vaccination 14 days prior to Visit 10 (6 months after study vaccination).
20. Receipt of live, attenuated vaccine 60 days prior to study enrollment, planned vaccination prior to completion of Visit 09 (Day 28 after study vaccination), or planned vaccination 14 days prior to Visit 10 (6 months after study vaccination).
21. History of Guillain-Barré Syndrome
22. Pregnant or lactating woman
23. Use of investigational agents within 30 days prior to study enrollment or planned use during the study period.
24. Donation of the equivalent of a unit of blood within 6 weeks prior to study enrollment, or during the first 5 weeks of study participation.
25. A member of the study team or their family member, to include investigators, research laboratory staff, clinical research staff.
26. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Dekker, MD, Principal Investigator — Stanford University; Stephen Quake, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: Yes
The NIH Human Immunology Project Consortium (HIPC) data repositories (ImmPORT) may store the results of the research assays results. Genetic data that is developed in this study may be made available to other researchers through the National Center for Biotechnology Information (NCBI) databases. Results from research assays will be labeled with a unique ID code and the volunteer identity (except for age) will not be disclosed.

REFERENCES:
- [Background] Lee J, Boutz DR, Chromikova V, Joyce MG, Vollmers C, Leung K, Horton AP, DeKosky BJ, Lee CH, Lavinder JJ, Murrin EM, Chrysostomou C, Hoi KH, Tsybovsky Y, Thomas PV, Druz A, Zhang B, Zhang Y, Wang L, Kong WP, Park D, Popova LI, Dekker CL, Davis MM, Carter CE, Ross TM, Ellington AD, Wilson PC, Marcotte EM, Mascola JR, Ippolito GC, Krammer F, Quake SR, Kwong PD, Georgiou G. Molecular-level analysis of the serum antibody repertoire in young adults before and after seasonal influenza vaccination. Nat Med. 2016 Dec;22(12):1456-1464. doi: 10.1038/nm.4224. Epub 2016 Nov 7. PMID 27820605
- [Derived] Horns F, Vollmers C, Dekker CL, Quake SR. Signatures of selection in the human antibody repertoire: Selective sweeps, competing subclones, and neutral drift. Proc Natl Acad Sci U S A. 2019 Jan 22;116(4):1261-1266. doi: 10.1073/pnas.1814213116. Epub 2019 Jan 8. PMID 30622180
- [Derived] de Bourcy CF, Angel CJ, Vollmers C, Dekker CL, Davis MM, Quake SR. Phylogenetic analysis of the human antibody repertoire reveals quantitative signatures of immune senescence and aging. Proc Natl Acad Sci U S A. 2017 Jan 31;114(5):1105-1110. doi: 10.1073/pnas.1617959114. Epub 2017 Jan 17. PMID 28096374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During spring and early summer (prior to June 30) of 2012, 11 participants were consented to participate. One participant was found to be ineligible and was therefore withdrawn prior to any interventions.
Groups:
- 2011-2012 Fluzone IIV3 (IM): 2011-2012 Fluzone IIV3 NDC No 49281-011-50
  2011-2012 Fluzone IIV3: This vaccine is given intramuscularly (IM)
Period: Overall Study
Arm/Group | 2011-2012 Fluzone IIV3 (IM)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants between the ages of 18-30
Arm/Group | 2011-2012 Fluzone IIV3 (IM)
Number analyzed (Participants) | 10
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 30 years old | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received Influenza Vaccine
Time Frame: Day 0 to 180 post-immunization
Population: 10 participants received the 2011-2012 Fluzone IIV3 vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | 2011-2012 Fluzone IIV3 (IM)
Number analyzed (Participants) | 10
Participants | 10

2. Secondary Outcome: Number of Participants With Related Adverse Events
Time Frame: Day 0 to 180 post-immunization
Population: Number of participants with related adverse events up to 180 days post immunization
Measure: Count of Participants; unit: Participants
Arm/Group | 2011-2012 Fluzone IIV3 (IM)
Number analyzed (Participants) | 10
Participants | 0

3. Other Pre Specified Outcome: Proteomic Analysis of Antibody CDR3 Regions at 10 Different Time Points Before and After Immunization.
Description: Proteomic analysis: Identification, production, and characterization of Influenza A specific antibodies and their CDRH3 amino-acid sequences.
Time Frame: Day -5 to 180 post-immunization
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 180 days post immunization
Arm/Group | 2011-2012 Fluzone IIV3 (IM)
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2011-2012 Fluzone IIV3 (IM) (N=10)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Pain in lumbosacral area
Upper respiratory infection (Infections and infestations) | 1 (1)
Abrasion LT upper leg (Skin and subcutaneous tissue disorders) | 1 (1) — Bike Accident

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No